CLINICAL TRIAL: NCT07043881
Title: Assessing Knowledge, Practices, Attitudes and Barriers of Puplic Population Regarding Helicobacter Pylori Infection in Upper Egypt: Cross- Sectional Study
Acronym: Hpylori/KAP
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Clinical Lecturer, Assiut University
Other Study IDs: 4-2025-300625
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Describe Current Practices in Hpylori Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess non medical population knowledge of H. pylori epidemiology, diagnostic methods, treatment guidelines, and complications.

Evaluate attitudes toward the importance of testing, eradication, and antibiotic resistance concerns.

Describe current practices in diagnosis, treatment regimens, and follow-up. Identify barriers (e.g., access to tests, cost, training) impacting management.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a gram-negative bacterium that colonizes the human stomach and is known for its role in the development of various gastrointestinal diseases. It is a major etiological factor in chronic peptic ulcer disease, which includes both gastric and duodenal ulcers.

The bacterium's ability to survive in the acidic environment of the stomach is facilitated by its production of urease, which neutralizes stomach acid. Chronic infection with H. pylori can lead to severe complications such as peptic ulcers, gastritis, and chronic indigestion (dyspepsia) making it a significant public health concern worldwide. It can lead to serious conditions such as stomach cancer (gastric adenocarcinoma) and mucosa-associated lymphoid tissue (MALT) lymphoma.

Helicobacter Pylori is one of the most common chronic infections that infect approximately 4.4 billion individuals worldwide. The area with the highest reported prevalence was reported in Africa (70.1%) while the lowest prevalence was reported in Switzerland (18.9%). The prevalence of HP shows large geographical variation with infection rates much higher in developing countries (in some areas > 85 %) than in Europe and North America (approximately 30%-40%). In various developing countries, more than 80% of the population is HP positive, even at young ages.

The significance of conducting research on H. pylori lies in its substantial burden on global health. Peptic ulcer disease and gastric cancer, both of which are associated with H. pylori infection, result in considerable morbidity and mortality.

Understanding the epidemiology, transmission dynamics, and pathogenic mechanisms of H. pylori is crucial for developing better prevention and treatment strategies. Additionally, research into antibiotic resistance patterns is essential for informing clinical practice and ensuring the continued efficacy of eradication regimens. Current research has extensively documented the global prevalence of H. pylori, with infection rates varying widely across different regions and populations.

Despite its widespread occurrence, there is a need to explore the knowledge and awareness of this infection within specific demographic segments, such as the urban population of Upper Egypt.

The level of awareness and knowledge about H. pylori in urban settings is crucial for public health initiatives, as it can inform targeted educational programs and interventions.

The urban population of the Upper Egypt, marked by diverse lifestyles and healthcare access, may exhibit unique patterns of awareness and knowledge regarding HP.

Factors such as cultural practices, dietary habits, and healthcare-seeking behavior can influence the prevalence of knowledge about the infection. Additionally, considering the rapid urbanization and lifestyle changes in Upper Egypt, exploring the awareness of H. pylori becomes increasingly relevant for developing effective preventive measures and promoting early detection.

ELIGIBILITY:
Inclusion Criteria:

* Non medical personnels.
* Age more than 18 years old e.g: patients, relatives of patients...etc.
* All persons who provided informed consent were included in this study.

Exclusion Criteria:

* All medical staff members

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Puplic population in Upper Egypt ( Assuit, Sohag, Minya, Qena, Luxor, Aswan) will answer validated, self-administered questionnaire (paper-based in Arabic).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Assess non medical population knowledge of H. pylori epidemiology, diagnostic methods, treatment guidelines, and complications. | one year
  Validated, self-administered questionnaire (paper-based in Arabic).